CLINICAL TRIAL: NCT06971432
Title: Comparison of the Effectiveness of Serratus Anterior Plane Block and Serratus Anterior Plane Block + Continuous Wound Infiltration With Catheter on Postoperative Pain After Minimally Invasive Cardiac Surgery
Brief Title: Serratus Anterior Plane Block and Serratus Anterior Plane Block + Continuous Wound Infiltration With Catheter
Acronym: MICS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Seda Kurtbeyoğlu, doctor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAPB / SAPB + LİA
Record Dates: First submitted 2025-05-04; First posted 2025-05-14 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Postoperative Pain; Minimal Invasive Cardiac Surgery
Keywords: minimal invasive cardiac surgery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Among the patients planned to undergo elective minimally invasive coronary bypass surgery, those who met the inclusion criteria were divided into two groups using the sealed envelope method by a researcher who would not be involved in any other phase of the study.
  After intubation and central vein cannulation were performed during the intraoperative period, the block method selected for the patient was applied.
  Patient data were recorded during the perioperative period.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group SAPB (Experimental): SAPB :Using ultrasound guidance, the needle is advanced in-plane at approximately 45° toward the fifth rib. For the superficial SAPB, the local anesthetic is injected anteriorly to the serratus anterior in the plane created with the latissimus dorsi muscle. The thoracodorsal artery runs in this plane, and while care should be taken not to puncture this vessel, the spread of the injectate around the vessel confirms the appropriate injection plane. For the deep SAPB, the local anesthetic is injected anteriorly to the rib and deep to the serratus anterior.
  Deep and superficial serratus anterior plane block (SAPB) will be performed at the level of the 5th rib. A total of 40 ml of 0.25% bupivacaine will be administered-20 ml into each compartment.
  All patients will routinely receive paracetamol 1 g four times daily. If the VAS score is 4 or higher, 100 mg of tramadol HCl will be administered.
  Interventions: Procedure: Group SAPB
- Group SAPB + LIA (Experimental): SAPB is applied similarly to the other group. Deep and superficial serratus anterior plane block (SAPB) will be performed at the level of the 5th rib. A total of 40 ml of 0.25% bupivacaine will be administered-20 ml into each compartment.At the end of the surgical procedure, while the incision line is still open, a catheter will be placed in the subcutaneous tissue, at the most lateral part of the incision. A 0.20% bupivacaine solution will be prepared and at the end of the operation, a 10 ml bolus will be administered, followed by a 2 ml/hour infusion for 48 hours.
  All patients will routinely receive paracetamol 1 g four times daily. If the VAS score is 4 or higher, 100 mg of tramadol HCl will be administered.
  Interventions: Procedure: Group SAPB + LIA

INTERVENTIONS:
Procedure: Group SAPB — Using ultrasound guidance, the needle is advanced in-plane at approximately 45° toward the fifth rib. For the superficial SAPB, the local anesthetic is injected anteriorly to the serratus anterior in the plane created with the latissimus dorsi muscle. The thoracodorsal artery runs in this plane, and while care should be taken not to puncture this vessel, the spread of the injectate around the vessel confirms the appropriate injection plane. For the deep SAPB, the local anesthetic is injected anteriorly to the rib and deep to the serratus anterior. Deep and superficial serratus anterior plane block (SAPB) will be performed at the level of the 5th rib. A total of 40 ml of 0.25% bupivacaine will be administered-20 ml into each compartment. All patients will routinely receive paracetamol 1 g four times daily. If the VAS score is 4 or higher, 100 mg of tramadol HCl will be administered.
  Arms: Group SAPB
Procedure: Group SAPB + LIA — SAPB is applied similarly to the other group.Deep and superficial serratus anterior plane block (SAPB) will be performed at the level of the 5th rib. A total of 40 ml of 0.25% bupivacaine will be administered-20 ml into each compartment.At the end of the surgical procedure, while the incision line is still open, a catheter will be placed in the subcutaneous tissue, at the most lateral part of the incision. A 0.20% bupivacaine solution will be prepared and at the end of the operation, a 10 ml bolus will be administered, followed by a 2 ml/hour infusion for 48 hours.
  All patients will routinely receive paracetamol 1 g four times daily. If the VAS score is 4 or higher, 100 mg of tramadol HCl will be administered.
  Arms: Group SAPB + LIA

SUMMARY:
A total of 46 patients scheduled to undergo elective coronary artery bypass surgery via a minimally invasive technique will be included in the study. In the preoperative period, patients will be randomly assigned into two groups using the sealed envelope method (SAPB / PECS II).

Upon arrival in the operating room, patients will undergo ECG and SpO₂ monitoring, followed by intra-arterial cannulation for continuous blood pressure monitoring. Anesthesia induction will be performed with 1 mg/kg lidocaine, 2-3 mg/kg propofol, 3 mcg/kg fentanyl, and 0.6 mg/kg rocuronium. Following endotracheal intubation, jugular vein cannulation will be performed.

Group 1:

Deep and superficial serratus anterior plane block (SAPB) will be performed at the level of the 5th rib. A total of 40 ml of 0.25% bupivacaine will be administered-20 ml into each compartment.

Group 2:

Deep and superficial serratus anterior plane block (SAPB) will be performed at the level of the 5th rib. A total of 40 ml of 0.25% bupivacaine will be administered-20 ml into each compartment.At the end of the surgical procedure, while the incision line is still open, a catheter will be placed in the subcutaneous tissue, at the most lateral part of the incision. A 0.20% bupivacaine solution will be prepared and at the end of the operation, a 10 ml bolus will be administered, followed by a 2 ml/hour infusion for 48 hours.

The following variables will be recorded: patient age, height, body weight, BMI, gender, type of analgesia administered, diagnosis, surgical procedure performed, any complications during or after the procedure, postoperative visual analogue scale (VAS) pain scores, additional postoperative analgesic use, patient satisfaction, postoperative nausea and vomiting, ICU length of stay, and total hospital length of stay.

All patients will routinely receive paracetamol 1 g four times daily. If the VAS score is 4 or higher, 100 mg of tramadol HCl will be administered.

DETAILED DESCRIPTION:
SAPB :Using ultrasound guidance, the needle is advanced in-plane at approximately 45° toward the fifth rib. For the superficial SAPB, the local anesthetic is injected anteriorly to the serratus anterior in the plane created with the latissimus dorsi muscle. The thoracodorsal artery runs in this plane, and while care should be taken not to puncture this vessel, the spread of the injectate around the vessel confirms the appropriate injection plane. For the deep SAPB, the local anesthetic is injected anteriorly to the rib and deep to the serratus anterior.

ELIGIBILITY:
Inclusion Criteria:

* Women and men aged 18-75,
* ASA I-II-III risk group,
* Body mass index between 18-35,
* who will undergo coronary artery bypass surgery with minimally invasive cardiac surgery method

Exclusion Criteria:

* Those under 18 and over 75
* Those with advanced comorbidities
* Those with ASA score IV
* Those with a history of bleeding diathesis and those using drugs that cause bleeding disorders
* Patients with an infection in the area where the block will be performed
* Patients who are allergic to the local anesthetic agent to be used
* Patients with a body mass index (BMI) under 18 and over 35 will be excluded from the study.

Withdrawal criteria:

* Patients who want to leave the study group
* Patients who develop surgical complications will be removed from the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 48 hours
  The patient will be visited at postoperative hours 0, 3, 6, 12, and 24, and their pain will be assessed. The patient will be asked to provide a number from 0 to 10 to rate the intensity of their pain, and the response will be recorded. A score of 0 indicates no pain, and 10 indicates unbearable, severe pain. Measurements will be taken four times:
  T4: 6th hour postoperatively
  T5: 12th hour postoperatively
  T6: 24th hour postoperatively
  T7: 48th hour postoperatively

SECONDARY OUTCOMES:
Heart Rate | 48 hours
  ECG monitoring was performed on the patient, and both rhythm and heart rate were observed. Heart rate was recorded as a numeric value per second. Measurements will be taken seven times:
  T1: Before induction
  T2: Within 5 minutes after the cardiopulmonary perfusion pump reaches full flow
  T3: Within 5 minutes after weaning from the cardiopulmonary perfusion pump
  T4: 6th hour postoperatively
  T5: 12th hour postoperatively
  T6: 24th hour postoperatively
  T7: 48th hour postoperatively
Mean Arterial Blood Pressure | 48 hours
  Intra-arterial cannulation and monitoring were established before induction. Mean arterial blood pressure was measured and recorded in mmHg. Measurements will be taken seven times:
  T1: Before induction
  T2: Within 5 minutes after the cardiopulmonary perfusion pump reaches full flow
  T3: Within 5 minutes after weaning from the cardiopulmonary perfusion pump
  T4: 6th hour postoperatively
  T5: 12th hour postoperatively
  T6: 24th hour postoperatively
  T7: 48th hour postoperatively
Oxygen Saturation | 48 hours
  Oxygen saturation was measured using a pulse oximeter on the second finger of the hand. It was recorded as a numeric value between 0 and 100. Measurements will be taken seven times:
  T1: Before induction
  T2: Within 5 minutes after the cardiopulmonary perfusion pump reaches full flow
  T3: Within 5 minutes after weaning from the cardiopulmonary perfusion pump
  T4: 6th hour postoperatively
  T5: 12th hour postoperatively
  T6: 24th hour postoperatively
  T7: 48th hour postoperatively
Additional Analgesics | 48 hours
  It will be assessed whether there is a need for additional analgesics within the first 24 hours. If additional analgesics are required, it will be recorded whether tramadol was administered. If it was, the number of times it was required and the dosage given will be noted. Assessments will be made at the following time points:
  T4: 6th hour postoperatively
  T5: 12th hour postoperatively
  T6: 24th hour postoperatively
  T7: 48th hour postoperatively
Nausea | 48 hours
  The patient will be interviewed and assessed for the frequency of opioid-related side effects during hospital visits. The patient will be visited at postoperative hours 6, 12, 24, and 48, and their nausea will be evaluated. The patient will be asked to rate the severity of their nausea on a scale from 0 to 10. A score of 0 indicates no nausea, while 10 indicates severe nausea.
Vomiting | 48 hours
  The patient will be interviewed and assessed for the frequency of opioid-related side effects during hospital visits. The patient will be visited at postoperative hours 6, 12, 24, and 48, and vomiting will be evaluated. If the patient has vomited, the number of episodes will be recorded. The total number of vomiting episodes within 48 hours will be documented.
Itching | 48 hours
  The patient will be interviewed and assessed for the frequency of opioid-related side effects during hospital visits. They will be evaluated at 6, 12, 24, and 48 hours postoperatively and asked whether they are experiencing pruritus. If present, the severity will be rated as mild, moderate, or severe.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jannati M, Attar A. Analgesia and sedation post-coronary artery bypass graft surgery: a review of the literature. Ther Clin Risk Manag. 2019 Jun 20;15:773-781. doi: 10.2147/TCRM.S195267. eCollection 2019. PMID 31417264
- [Result] Ekinci M, Ciftci B, Golboyu BE, Demiraran Y, Bayrak Y, Tulgar S. A Randomized Trial to Compare Serratus Anterior Plane Block and Erector Spinae Plane Block for Pain Management Following Thoracoscopic Surgery. Pain Med. 2020 Jun 1;21(6):1248-1254. doi: 10.1093/pm/pnaa101. PMID 32417925
- [Result] Thompson C, French DG, Costache I. Pain management within an enhanced recovery program after thoracic surgery. J Thorac Dis. 2018 Nov;10(Suppl 32):S3773-S3780. doi: 10.21037/jtd.2018.09.112. PMID 30505564
- [Result] Berthoud V, Ellouze O, Nguyen M, Konstantinou M, Aho S, Malapert G, Girard C, Guinot PG, Bouchot O, Bouhemad B. Serratus anterior plane block for minimal invasive heart surgery. BMC Anesthesiol. 2018 Oct 20;18(1):144. doi: 10.1186/s12871-018-0614-5. PMID 30340525
- [Result] Saikat S, Shweta S, Somalia M, Dibyendu K, Sushan M. Comparative efficacy of serratus anterior plane block (SAPB) and fentanyl for postoperative pain management and stress response in patients undergoing minimally invasive cardiac surgery (MICS). Ann Card Anaesth. 2023 Jul-Sep;26(3):268-273. doi: 10.4103/aca.aca_91_22. PMID 37470524